CLINICAL TRIAL: NCT00334815
Title: A Pilot Trial of Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Docetaxel and the Addition of Bevacizumab (NSC-704865) in Three Cohorts of Patients With Inoperable Locally Advanced Stage III Non-small Cell Lung Cancer
Brief Title: Combination Chemotherapy, Radiation Therapy, and Bevacizumab in Treating Patients With Newly Diagnosed Stage III Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01097; NCI-2009-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0533; CDR0000472907; S0533 (Other: SWOG); S0533 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Lung Adenocarcinoma; Lung Adenosquamous Carcinoma; Lung Large Cell Carcinoma; Lung Squamous Cell Carcinoma; Minimally Invasive Lung Adenocarcinoma; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Radiotherapy; Radiation

ARMS (3):
- Group 1 (cisplatin, etoposide, radiotherapy) (Experimental): Patients receive cisplatin IV over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Patients undergo concurrent thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Etoposide; Biological: Filgrastim; Biological: Pegfilgrastim; Radiation: Radiation Therapy
- Group 2 (cisplatin, etoposide, radiotherapy, bevacizumab) (Experimental): Patients receive cisplatin, etoposide, and thoracic radiotherapy as in group 1. Patients also receive bevacizumab IV over 30-90 minutes on days 15, 36, and 57.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Docetaxel; Drug: Etoposide; Biological: Filgrastim; Biological: Pegfilgrastim; Radiation: Radiation Therapy
- Group 3 (cisplatin, etoposide, radiotherapy, bevacizumab) (Experimental): Patients receive cisplatin, etoposide, and thoracic radiotherapy as in group 1. Patients also receive bevacizumab IV over 30-90 minutes on days 1, 22, and 43.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Docetaxel; Drug: Etoposide; Biological: Filgrastim; Biological: Pegfilgrastim; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Group 2 (cisplatin, etoposide, radiotherapy, bevacizumab); Group 3 (cisplatin, etoposide, radiotherapy, bevacizumab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Radiation: Radiation Therapy — Undergo thoracic radiotherapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This clinical trial studies combination chemotherapy, radiation therapy, and bevacizumab in treating patients with newly diagnosed stage III non-small cell lung cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as cisplatin, etoposide, and docetaxel, work in different ways to stop the growth of [cancer/tumor] cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving more than one drug (combination chemotherapy) together with radiation therapy and bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency and severity of toxic effects of induction therapy comprising cisplatin, etoposide, and radiotherapy with or without bevacizumab followed by consolidation therapy comprising docetaxel and bevacizumab, in terms of grade 4 or 5 hemorrhage, in patients with newly diagnosed, unresectable, stage III non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. Determine progression-free and overall survival of patients treated with these regimens.

II. Determine response (confirmed, unconfirmed, partial, and complete) in patients with measurable disease treated with these regimens.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to risk (high* vs low).

NOTE: *High-risk stratum closed to accrual as of 2/20/09.

INDUCTION THERAPY: Patients in each stratum are assigned to 1 of 3 sequential treatment groups.

GROUP 1: Patients receive cisplatin intravenously (IV) over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Patients undergo concurrent thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.

GROUP 2: Patients receive cisplatin, etoposide, and thoracic radiotherapy as in group 1. Patients also receive bevacizumab IV over 30-90 minutes on days 15, 36, and 57.

GROUP 3: Patients receive cisplatin, etoposide, and thoracic radiotherapy as in group 1. Patients also receive bevacizumab IV over 30-90 minutes on days 1, 22, and 43.

CONSOLIDATION CHEMOTHERAPY: Beginning 3-6 weeks after completion of induction therapy, all patients receive consolidation chemotherapy comprising docetaxel IV over 1 hour and bevacizumab IV over 30-90 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 2 and continuing until blood counts recover OR pegfilgrastim SC once on day 2.

Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed single, primary, bronchogenic, non-small cell lung cancer (NSCLC)

  * Newly diagnosed disease
  * Unresectable disease
  * No more than 1 parenchymal lesions on same or opposite sides of the lungs
* Meets 1 of the following stage criteria:

  * Stage IIIA (N2) disease meeting the following criteria:

    * N2 mediastinal lymph nodes must be multiple and/or bulky on CT scan or x-ray so that the patient is not a candidate for induction chemotherapy or chemoradiotherapy followed by surgical resection
    * N2 status must be documented by ≥ 1 of the following methods:

      * Histologically or cytologically confirmed N2 disease by exploratory thoracotomy, thoracoscopy, mediastinoscopy, mediastinotomy, Chamberlain procedure, Wang needle biopsy (WNB), fine needle aspiration (FNA) under bronchoscopic or CT guidance, or any other method
      * Node positive by fludeoxyglucose-positron emission tomography (FDG-PET) scan
      * Nodes > 3 cm on CT scan
      * Paralyzed left true vocal cord with separate left lung primary distinct from anterior-posterior window nodes on CT scan
  * Stage IIIB disease meeting ≥ 1 of the following criteria:

    * Histologically or radiographically confirmed positive N3 nodes*, documented by ≥ 1 of the following methods:

      * FNA, core needle biopsy (CNB), or excisional biopsy of supraclavicular N3 nodes
      * Biopsy of contralateral mediastinal N3 nodes by mediastinoscopy, mediastinotomy, or thoracotomy
      * FNA, CNB, or WNB under CT or bronchoscopic fluoroscopic guidance of enlarged contralateral N3 mediastinal nodes
      * Contralateral mediastinal nodes > 3 cm on CT scan
      * Node positivity by FDG-PET scan
      * Right-sided primary with paralyzed left true vocal cord
    * T4 lesions of any size that invade the mediastinum, heart, great vessels, trachea, esophagus, vertebral body, or carina, documented by ≥ 1 of the following methods:

      * Written documentation of type of T4 extent if patient had a prior exploratory thoracotomy or thoracoscopy
      * T4 involvement of the trachea or carina by direct bronchoscopic visualization
      * T4 involvement of the heart, esophagus, aorta, or vertebral body by CT scan, MRI, or transesophageal ultrasound
      * T4 involvement of the mediastinum by CT scan or MRI if, in the absence of the above organ involvement, there is soft tissue extension directly into the mediastinal space**
* Meets 1 of the following risk criteria:

  * Low risk disease, meeting the following criteria:

    * Non-squamous cell NSCLC, including adenocarcinoma, bronchoalveolar cell carcinoma, or large cell carcinoma

      * If mixed histology, the squamous cell carcinoma component must be < 50%
      * Histology or cytology from involved mediastinal or supraclavicular lymph nodes allowed if a separate distal primary lesion is clearly evident on radiographs (i.e., second biopsy not required)
    * No primary tumor with cavitation and/or tumor within 1 cm of a major vessel
    * No hemoptysis (i.e., bright red blood ≥ ½ teaspoon) in the past 28 days
  * High-risk* disease, meeting ≥ 1 of the following criteria:

    * Squamous cell NSCLC

      * If mixed histology, the squamous cell component must be ≥ 50%
    * Tumor with any histology that has cavitation or is located within 1 cm of a major vessel

      * No aortic involvement
    * Any histology and hemoptysis (i.e., bright red blood ≥ ½ teaspoon) within past 28 days
* Measurable or nonmeasurable disease by CT scan or MRI

  * Pleural effusions, ascites, and laboratory parameters are not acceptable as the only evidence of disease
* No pleural effusion except for small pleural effusion visible on CT scan or MRI alone
* No pericardial effusions
* No metastatic disease involving the contralateral chest, liver, or adrenals confirmed by CT scan of the upper abdomen or by chest CT scan with complete liver and adrenals in the report
* Patients must be offered participation in SWOG-S9925 (Lung Cancer Specimen Repository Protocol)
* No brain metastases by CT scan or MRI
* No evidence of cavitation
* Creatinine normal
* Creatinine clearance ≥ 50 mL/min
* FEV_1 ≥ 2.0 liters OR predicted FEV_1 of the contralateral lung > 800 mL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Urine protein: creatinine ratio ≤ 0.5 by urinalysis OR urine protein < 1,000 mg by 24-hour urine collection
* INR < 1.5
* Zubrod performance status 0-1
* No sensory neuropathy > grade 1
* No cerebrovascular accident within the past 6 months
* No myocardial infarction or unstable angina within the past 6 months
* No uncontrolled hypertension
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No pathologic condition other than lung cancer that carries a high risk of bleeding
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No serious, nonhealing wound, ulcer, or bone fracture
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer for which the patient is currently in complete remission, or other cancer for which the patient has been disease-free for 5 years
* Not pregnant or nursing

  * No nursing during and for ≥ 6 months after the last dose of bevacizumab
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after the last dose of bevacizumab
* Must have pre-treatment simulation demonstrating a V20 ≤ 35% with planned radiation dose of 6,480 cGy
* No prior surgical resection

  * Prior exploratory thoracotomy, mediastinoscopy, excisional biopsy, or similar surgery allowed for diagnosing, staging, or determining potential resectability of lung tumor
* No prior chemotherapy or radiotherapy for lung cancer
* No prior radiotherapy to the neck or thorax
* At least 4 weeks since prior thoracic or other major surgery (excluding mediastinoscopy) and recovered
* More than 7 days since prior FNA, CNB, or mediastinoscopy
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, or biologic agents
* No other concurrent investigational drugs
* No concurrent major surgical procedures
* No concurrent full-dose anticoagulants (e.g., low-molecular weight and unfractionated heparin or warfarin)

  * Low-dose warfarin (i.e., 1 mg) is allowed to prevent clotting of an infusaport or central line
* No concurrent brachytherapy, radiopharmaceuticals, high linear energy transfer radiation (i.e., fast neutrons), particle therapy (i.e., protons, carbon, or helium), and/or altered fractionation schemes
* No concurrent intensity-modulated radiotherapy
* No concurrent prophylactic contralateral hilar or supraclavicular lymph node radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06-15 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette J Wozniak, Principal Investigator — SWOG Cancer Research Network
Locations (63):
- United States (63):
  - Providence Hospital, Mobile, Alabama
  - Saint Bernards Regional Medical Center, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Roper Hospital, Charleston, South Carolina
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Risk Patient Stratum: Patients with non-squamous histology, a primary tumor with no cavitation and not within 1 cm of a major blood vessel, and no history of hemoptysis.
  Treatment received was cisplatin IV over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Patients undergo concurrent thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.
  cisplatin: Given IV
  etoposide: Given IV
  radiation therapy: Undergo thoracic radiotherapy
  docetaxel: Given IV
  filgrastim: Given SC
  pegfilgrastim: Given SC
- High Risk Patient Stratum: Patients with at least one of the following characteristics: squamous histology, a primary tumor with cavitation or within 1 cm of a major blood vessel, a history of hemoptysis.
  Treatment received was cisplatin IV over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Patients undergo concurrent thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.
  cisplatin: Given IV
  etoposide: Given IV
  radiation therapy: Undergo thoracic radiotherapy
  docetaxel: Given IV
  filgrastim: Given SC
  pegfilgrastim: Given SC
Period: Overall Study
Arm/Group | Low Risk Patient Stratum | High Risk Patient Stratum
Started | 16 | 13
Completed | 9 | 3
Not Completed | 7 | 10
Not completed — Adverse Event | 3 | 2
Not completed — Death | 0 | 2
Not completed — Progression | 1 | 0
Not completed — ineligible | 1 | 1
Not completed — patient refused treatment | 0 | 1
Not completed — Physician Decision | 2 | 4

BASELINE CHARACTERISTICS:
Population: All eligible patients who received protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Patient Stratum | High Risk Patient Stratum | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Continuous [Median (Full Range); unit: years] | 54.5 [32.4 to 70.3] | 63.4 [51.1 to 77.2] | 60.5 [32.4 to 77.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to one year
Population: All eligible patients, both low-risk and high-risk strata combined, who received protocol therapy.
Measure: Number; unit: Participants
Arm/Group | Concurrent Chemotherapy and Radiotherapy | Consolidation Therapy With Docetaxel and Bevacizumab.
Number analyzed (Participants) | 26 | 21
Participants
  Acidosis (metabolic or respiratory) | 0 | 1
  Arthritis (non-septic) | 0 | 1
  Calcium, serum-low (hypocalcemia) | 0 | 1
  Carbon monoxide diffusion capacity (DL(co)) | 1 | 0
  Creatinine | 1 | 0
  Dehydration | 1 | 0
  Dyspnea (shortness of breath) | 1 | 1
  Esophagitis | 2 | 0
  FEV(1) | 1 | 0
  Febrile neutropenia | 3 | 0
  Glucose, serum-high (hyperglycemia) | 1 | 0
  Hemoglobin | 2 | 2
  Hemorrhage, Respiratory tract NOS | 0 | 1
  Hemorrhage, GI - Peritoneal cavity | 0 | 1
  Hemorrhage, pulmonary/upper respiratory - Lung | 0 | 1
  Hypotension | 1 | 0
  Hypoxia | 0 | 1
  INR (of prothrombin time) | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Nose | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 0
  Leukocytes (total WBC) | 6 | 0
  Lymphopenia | 2 | 3
  Muscle weakness, not d/t neuropathy - body/general | 1 | 1
  Nausea | 2 | 0
  Neutrophils/granulocytes (ANC/AGC) | 10 | 0
  Pain - Chest wall | 1 | 0
  Pain - Chest/thorax NOS | 1 | 0
  Pain - Head/headache | 1 | 0
  Pain - Joint | 0 | 1
  Pain - Neck | 1 | 0
  Pain - Throat/pharynx/larynx | 1 | 0
  Platelets | 2 | 0
  Pneumonitis/pulmonary infiltrates | 1 | 2
  Potassium, serum-low (hypokalemia) | 3 | 1
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1
  Rash/desquamation | 1 | 0
  Rash: dermatitis associated w/radiation | 1 | 0
  Sodium, serum-low (hyponatremia) | 1 | 0
  Weight loss | 0 | 1

2. Secondary Outcome: Progression-free Survival
Description: From date of registration to time of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: Disease assessments were performed every 10 weeks as long as the patient remained on protocol treatment, up to 4 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Low Risk Patient Stratum | High Risk Patient Stratum
Number analyzed (Participants) | 15 | 11
Months | 38 [23 to 46] | 15 [5 to 17]

3. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Every week, up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Low Risk Patient Stratum | High Risk Patient Stratum
Number analyzed (Participants) | 15 | 11
Months | 46 [26 to 51] | 17 [5 to 18]

4. Secondary Outcome: Response Rate (Confirmed or Unconfirmed Partial Response)
Description: Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions.
Time Frame: Response assessment occured at the end of CRT and docetaxel/bevacizumab and then every 2-3 months for 2 years and then every 6 months until 4 years after the initial registration
Population: Only patients with measurable disease at baseline were included in the analysis of response. Among 15 patients on the Low Risk stratum, 14 had measureable disease at baseline. Among 11 patients on the High Risk stratum, 10 had measureable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Risk Patient Stratum | High Risk Patient Stratum
Number analyzed (Participants) | 14 | 10
percentage of participants | 64 [35 to 87] | 70 [35 to 93]

ADVERSE EVENTS:
Time Frame: Up to one year.
Groups:
- Concurrent Chemotherapy and Radiotherapy: All eligible patients, both low-risk and high-risk strata combined, who received concurrent chemotherapy and radiotherapy.
- Consolidation Therapy With Docetaxel and Bevacizumab: All eligible patients, both low-risk and high-risk strata combined, who received consolidation therapy with Docetaxel and Bevacizumab.
Arm/Group | Concurrent Chemotherapy and Radiotherapy | Consolidation Therapy With Docetaxel and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/26 | 3/21
Other Adverse Events (participants affected / at risk) | 26/26 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Chemotherapy and Radiotherapy (N=26) | Consolidation Therapy With Docetaxel and Bevacizumab (N=21)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Hemorrhage, GI - Peritoneal cavity (Gastrointestinal disorders) | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Chemotherapy and Radiotherapy (N=26) | Consolidation Therapy With Docetaxel and Bevacizumab (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Hemoglobin (Blood and lymphatic system disorders) | 9 | 8
Vision-blurred vision (Eye disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 10 | 1
Esophagitis (Gastrointestinal disorders) | 12 | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 17 | 4
Pain - Esophagus (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 9 | 3
Edema: limb (General disorders) | 2 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21 | 10
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3 | 0
Pain - Chest/thorax NOS (General disorders) | 4 | 4
Rigors/chills (General disorders) | 3 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2 | 0
Rash: dermatitis associated w/Chemoradiation (Injury, poisoning and procedural complications) | 2 | 2
Rash: dermatitis associated w/radiation (Injury, poisoning and procedural complications) | 4 | 0
Creatinine (Investigations) | 2 | 0
Leukocytes (total WBC) (Investigations) | 9 | 2
Lymphopenia (Investigations) | 6 | 3
Metabolic/Laboratory-Other (Investigations) | 0 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 14 | 0
Platelets (Investigations) | 10 | 5
Weight loss (Investigations) | 6 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 8 | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 | 6
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 1
Neuropathy: sensory (Nervous system disorders) | 2 | 5
Pain - Head/headache (Nervous system disorders) | 5 | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 3 | 1
Confusion (Psychiatric disorders) | 2 | 0
Renal/Genitourinary-Other (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 | 2
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less